CLINICAL TRIAL: NCT03764501
Title: Image Fusion System for 3D Preoperative Planning in the Osteosynthesis and Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokyo Medical University (Other)
Responsible Party: Principal Investigator, Yuichi Yoshii, Associate Professor, Department of Orthopaedic Surgery, Tokyo Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-19
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Fractures, Bone; Fracture Malunion, Bone
MeSH Terms: conditions — Fractures, Bone; Fractures, Malunited

STUDY DESIGN:
Intervention Model Description: Image fusion group will utilize 3D preoperative planning and image fusion system. Control group will utilize only 3D preoperative planning.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Image fusion group (Image fusion) (Active Comparator): Use image fusion system during surgery (Image fusion, ZedTrauma, LEXI Co., Ltd.)
  Interventions: Device: Image fusion system
- Control group (ZedTrauma) (No Intervention): only use 3D preoperative planning (Zed Trauma, LEXI Co., Ltd.)

INTERVENTIONS:
Device: Image fusion system — Image fusion system for the 3D preoperative planning
  Arms: Image fusion group (Image fusion)

SUMMARY:
Utility of image fusion system for the fracture and fracture malunion management will be evaluated.

DETAILED DESCRIPTION:
The fracture and malunion patients need osteosynthesis or osteotomy will be recruited. Image fusion group utilizes 3D preoperative planning and image fusion system. Control group utilizes only 3D preoperative planning. The age, sex, and fracture types will be matched between groups. In both groups, 3D preoperative planning will be performed in order to determine reduction, placement and choices of implants. In the image fusion group, the outline of planned image will be displayed on the monitor overlapping with fluoroscopy image during surgery. Reductions, implant choices/positions, and clinical outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Fracture paitents need osteosynthesis

Exclusion Criteria:

* Fracture patients under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction accuracy | 1month after the surgery
  Reproducibility of the reduction shape will be measured.
Implant placement | 1month after the surgery
  Reproducibility of the implant placement will be evaluated.
Implant choices | 1month after the surgery
  Reproducibility of the implant choices will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo Medical University Ibaraki Medical Center, Ami, Ibaraki, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoshii Y, Ogawa T, Hara Y, Totoki Y, Ishii T. An image fusion system for corrective osteotomy of distal radius malunion. Biomed Eng Online. 2021 Jun 30;20(1):66. doi: 10.1186/s12938-021-00901-8. PMID 34193171
- [Derived] Yoshii Y, Totoki Y, Sashida S, Sakai S, Ishii T. Utility of an image fusion system for 3D preoperative planning and fluoroscopy in the osteosynthesis of distal radius fractures. J Orthop Surg Res. 2019 Nov 6;14(1):342. doi: 10.1186/s13018-019-1370-z. PMID 31694677